CLINICAL TRIAL: NCT01434095
Title: Microperimetric Evaluation After Half-dose Photodynamic Therapy for Chronic Central Serous Chorioretinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Surugadai Nihon University Hospital (Other)
Collaborators: Teikyo University (Other)
Responsible Party: Principal Investigator, Kyoko Fujita, Dr. Kyoko Fujita, MD, PhD, Surugadai Nihon University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 81004
Record Dates: First submitted 2011-09-13; First posted 2011-09-14 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Chronic Central Serous Chorioretinopathy
Keywords: microperimetry; fixation point; retinal sensitivity; photodynamic therapy; chronic central serous chorioretinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- half-dose PDT(photodynamic therapy) (Active Comparator): The study include single arm; treated group, and no control group was included.
  Interventions: Procedure: half-dose photodynamic therapy

INTERVENTIONS:
Procedure: half-dose photodynamic therapy — photodynamic therapy (PDT) was performed using 3 mg/m2 body surface area of verteporfin (Visudyne, Novartis AG, Bülach, Switzerland) which is one-half the conventional dose of verteporfin. The verteporfin was infused over a 10 minute period followed by the delivery of 50 J/cm2 from a 689-nm laser system (Carl Zeiss, Dublin, CA) over an 83-second exposure time.

SUMMARY:
A half-dose photodynamic therapy, a relative new treatment, has been widely performed to treat central serous chorioretinopathy.

The researchers aimed to investigate whether the therapy improved the patient's visual acuity as well as the retinal sensitivity. The researchers also investigate which clinical factors, if any, were associated with the results; visual acuity or retinal sensitivity after the treatment.

DETAILED DESCRIPTION:
The best-corrected visual acuity (BCVA), macular sensitivity, and fixation stability were evaluated at the baseline and at 1, 3, 6, and 12 months after the half-dose photodynamic therapy. The macular sensitivity and fixation stability were determined by MP-1 microperimetry (Nidek, Vigonza, Italy). The researchers analysed whether the BCVA and retinal sensitivity significantly improved or not. And if yes, the researchers were interested at which period after treatment the significant improvement was found. Also, the researchers investigated which improved first, BCVA or retinal sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* the presence of subretinal fluid involving the fovea in the Optical coherence tomographic (OCT) images
* a serous retinal detachment of at least 6 months duration.

Exclusion Criteria:

* evidence of a choroidal neovascularization (CNV), polypoidal choroidal vasculopathy, or other maculopathy documented by fluorescein angiography or Indocyanine green angiography

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
best corrected visual acuity | one year

SECONDARY OUTCOMES:
retinal sensitivity | one year

CONTACTS AND LOCATIONS:
Overall Officials: Kyoko Fujita, MD, PhD, Principal Investigator — Department of Ophthalmology, Surugadai Nihon University Hospital
Locations (1):
- Department of Ophthalmology, Surugadai Nihon University Hospital, Chiyoda-ku, Tokyo, Japan

REFERENCES:
- [Derived] Fujita K, Shinoda K, Imamura Y, Matsumoto CS, Mizutani Y, Mizota A, Yuzawa M. Correlation of integrity of cone outer segment tips line with retinal sensitivity after half-dose photodynamic therapy for chronic central serous chorioretinopathy. Am J Ophthalmol. 2012 Sep;154(3):579-85. doi: 10.1016/j.ajo.2012.03.043. Epub 2012 Jul 20. PMID 22818904